CLINICAL TRIAL: NCT07096843
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Efficacy of Budoprutug (TNT119) in Subjects With Primary Membranous Nephropathy (PMN)
Brief Title: A Phase 2 Study of Budoprutug in Subjects With Primary Membranous Nephropathy
Acronym: PrisMN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Climb Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNT119-PMN-201
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Primary Membranous Nephropathy
Keywords: PMN; Anti-CD19; PrisMN

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Dose Level A (Experimental)
  Interventions: Drug: budoprutug
- Cohort 2: Dose Level B (Experimental)
  Interventions: Drug: budoprutug
- Cohort 3: Dose Level C (Experimental)
  Interventions: Drug: budoprutug

INTERVENTIONS:
Drug: budoprutug — Single IV dose of study product on Day 1, Day 15, Day 169 and Day 183
  Other Names: TNT119

SUMMARY:
To evaluate the safety and tolerability of three dose regimens of budoprutug in subjects with PMN

DETAILED DESCRIPTION:
Budoprutug is a humanized, immunoglobulin (Ig) G1 monoclonal antibody that selectively binds to CD19 and is projected to deplete targeted cells through antibody-dependent cellular cytotoxicity (ADCC). This Phase 2, open-label, multicenter study evaluates the safety, pharmacodynamics, and preliminary efficacy of three intravenous dose regimens of budoprutug in adult subjects with primary membranous nephropathy (PMN) who are anti-PLA2R antibody positive and have persistent proteinuria despite optimized RAAS inhibition. Approximately 45 subjects will be enrolled across three sequential dose cohorts, each receiving a single IV dose of budoprutug on Day 1, Day 15, Day 169 and Day 183. Subjects will be followed through Week 48, with extended follow-up for B-cell recovery as needed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PMN with positive anti-PLA2R antibodies
* CD19+ B cell count ≥40 cells/μL
* UPCR ≥2.0 g/g
* eGFR ≥40 mL/min/1.73 m²
* Stable RAAS inhibitor therapy
* Blood pressure <150/90 mmHg at baseline
* Adequate hematologic, hepatic, and renal function
* Willing to use effective contraception (both sexes)
* Other inclusion criteria may apply

Exclusion Criteria:

* Secondary Membranous Nephropathy
* Rapidly progressive glomerulonephritis or other glomerulopathies
* Prior B cell-depleting therapy within 24 weeks
* Recent use of immunosuppressants
* Active or high-risk infections
* History of malignancy
* Pregnancy or breastfeeding
* Recent major surgery or hospitalization
* Other exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to Week 48
  Number of participants experiencing TEAEs, graded per NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Change in total B Cell Count | Up to Week 48
  Absolute and % change in total number of peripheral B cells over time.
Change in Anti-PLA2R Antibodies | Up to Week 48
  Change from Baseline in anti-PLA2R antibody titers over time.
Complete Remission Rate | Week 48
  Proportion of subjects who achieve complete remission at Week 48.
Complete or Partial Remission Rate | Week 48
  Proportion of subjects who achieve complete or partial remission at Week 48.
Change in Proteinuria | Up to Week 48
  Change from Baseline in proteinuria (measured via urine protein-creatinine ratio, UPCR) over time.
Change in UACR | Up to Week 48
  Change in urine albumin-to-creatinine ratio over time.
Change in eGFR | Up to Week 48
  Change from Baseline in eGFR over time.
Area Under the Curve (AUC) | Up to Week 48
  Measurement of the area under the drug concentration-time curve.
Maximum Observed Plasma Concentration (Cmax) | Up to Week 48
  Measurement of the maximum observed plasma concentration.
Time to Maximum Observed Concentration (Tmax) | Up to Week 48
  Measurement of the time to maximum observed concentration.
Terminal Half-Life (T1/2) | Up to Week 48
  Measurement of the terminal half-life in days.
Apparent Clearance (CL/F) | Up to Week 48
  Measurement of the apparent clearance in L/hour.
Volume of Distribution (Vd) | Up to Week 48
  Measurement of the volume of distribution in liters.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (8):
  - Climb Bio Investigative Site #110, Denver, Colorado
  - Climb Bio Investigative Site #105, Orlando, Florida
  - Climb Bio Investigative Site #108, Atlanta, Georgia
  - Climb Bio Investigative Site #106, Indianapolis, Indiana
  - Climb Bio Investigative Site #101, Clifton Park, New York
  - Climb Bio Investigative Site #102, Philadelphia, Pennsylvania
  - Climb Bio Investigative Site #103, El Paso, Texas
  - Climb Bio Investigative Site #104, Sherman, Texas
- Argentina (6):
  - Climb Bio Investigative Site# 602, Buenos Aires
  - Climb Bio Investigative Site# 603, Buenos Aires
  - Climb Bio Investigative Site #601, CABA
  - Climb Bio Investigative Site #604, CABA
  - Climb Bio Investigative Site #605, Córdoba
  - Climb Bio Investigative Site #606, Santa Fe
- Brazil (6):
  - Climb Bio Investigative Site #502, Belo Horizonte
  - Climb Bio Investigative Site #505, Minas Gerais
  - Climb Bio Investigative Site #506, Pernambuco
  - Climb Bio Investigative Site #501, Porto Alegre
  - Climb Bio Investigative Site #503, São Paulo
  - Climb Bio Investigative Site #504, São Paulo
- Chile (3):
  - Climb Bio Investigative Site #702, Santiago
  - Climb Bio Investigative Site #701, Temuco
  - Climb Bio Investigative Site# 703, Valdivia
- Georgia (3):
  - Climb Bio Investigative Site #903, Tbilisi
  - Climb Bio Investigative Site #902, Tbilisi
  - Climb Bio Investigative Site #901, Tbilisi
- Taiwan (5):
  - Climb Bio Investigative Site #204, Taichung
  - Climb Bio Investigative Site# 202, Taipei
  - Climb Bio Investigative Site# 201, Taipei
  - Climb Bio Investigative Site #205, Taipei
  - Climb Bio Investigative Site# 203, Taipei
- Ukraine (5):
  - Climb Bio Investigative Site #803, Ivano-Frankivsk
  - Climb Bio Investigative Site# 801, Kyiv
  - Climb Bio Investigative Site #805, Kyiv
  - Climb Bio Investigative Site #804, Rivne
  - Climb Bio Investigative Site #802, Ternopil

IPD SHARING:
Plan to Share IPD: No